CLINICAL TRIAL: NCT00404989
Title: Antiretroviral Pregnancy Registry
Brief Title: Antiretroviral Pregnancy Registry (APR): Multi-sponsor Registry to Detect Any Major Teratogenic Effect Involving Any of the Registry Drugs When Administered to Pregnant People.
Acronym: APR
Status: Recruiting | Type: Observational
Sponsor: Syneos Health (Other)
Collaborators: AbbVie (Industry); Alvogen Inc. (Unknown); Amneal Pharmaceuticals, LLC (Industry); Apotex Corp. (Unknown); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); Cipla Ltd. (Industry); Dr. Reddy's Laboratories Limited (Industry); Gilead Sciences (Industry); Hetero Labs (Unknown); Hikma Pharmaceuticals LLC (Industry); i3 Pharmaceuticals, LLC (Unknown); Janssen Scientific Affairs, LLC (Industry); Lannett Company, Inc. (Industry); Laurus Labs Limited (Unknown); Lupin Pharmaceuticals, Inc. (Industry); Macleods Pharmaceuticals Ltd (Industry); Merck Sharp & Dohme LLC (Industry); Mylan Laboratories (Industry); Pharmascience Inc. (Industry); Qilu Pharmaceutical Co., Ltd. (Industry); Sigmapharm Laboratories (Unknown); Strides Pharma Science Limited (Unknown); Teva Pharmaceuticals USA (Industry); ViiV Healthcare (Industry); Yung Shin Pharm. Ind. Co., Ltd. (Industry); Zydus Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: APR; NCT01137981 (obsolete NCT alias)
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections; Hepatitis B
Keywords: HIV; HBV; Hepatitis; Pregnancy; Registry
MeSH Terms: conditions — HIV Infections; Hepatitis B; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the Antiretroviral Pregnancy Registry (Registry) is to detect any major teratogenic effect involving any of the Registry drugs when administered to pregnant people. Registration is voluntary and confidential with information obtained from the health care provider. A Registry-assigned identifier allows for follow-up capability. Information on subjects is provided to the Registry prospectively (prior to the outcome of pregnancy being known) through their health care provider, with follow-up obtained from the health care provider after the outcome is determined. Providers are strongly urged to enroll their patients as early in pregnancy as possible to maximize the validity of the data. In addition, the Registry is very interested in assembling a group of providers who are willing to make a commitment to report all of their site's antiretroviral pregnancy exposures to the Registry, thereby assuring all cases can be considered prospective. Providers are encouraged to contact the Registry for more information about this group. The Registry is informed in its analysis by other data, for example, retrospective reports and clinical studies.

Given the increasing number of medications and more aggressive approach to therapy, more HIV- and hepatitis B-infected people may be treated during pregnancy or become pregnant while under treatment. The paucity of data on use and infant outcomes of antiretroviral therapies during pregnancy makes this Registry an essential component of the ongoing program of epidemiologic studies of the safety of these therapies.

Each year the Registry has enrolled approximately 1300-1700 pregnant people in the US exposed to antiretroviral drugs. This number represents approximately 15% of the 8,700 HIV positive people who give birth to live infants annually in the US.

DETAILED DESCRIPTION:
The following antiretroviral drugs are followed by the Antiretroviral Pregnancy Registry (APR, Registry) to detect any major teratogenic effect when administered to pregnant people: abacavir (ZIAGEN®, ABC), abacavir/lamivudine (EPZICOM®, KIVEXA®, EPZ), abacavir/lamivudine/zidovudine (TRIZIVIR®, TZV), abacavir/dolutegravir/lamivudine (TRIUMEQ®, TRI), adefovir dipivoxil (HEPSERA®, ADV), amprenavir (AGENERASE®, APV), atazanavir (REYATAZ®, ATV), atazanavir/cobicistat (EVOTAZ®, EVO), bictegravir/emtricitabine/tenofovir alafenamide (BIKTARVY®, B/F/TAF), cabotegravir (VOCABRIA®, CABENUVA®, APRETUDE®, CAB), cobicistat (TYBOST®, COBI), darunavir (PREZISTA®, DRV), darunavir/cobicistat (PREZCOBIX™, REZOLSTA™, PCX), darunavir/cobicistat/emtricitabine/tenofovir alafenamide (SYMTUZA®, DCF TAF ), delavirdine mesylate (RESCRIPTOR®, DLV), didanosine (VIDEX®, VIDEX® EC, ddI), dolutegravir (TIVICAY®, DTG), dolutegravir/lamivudine (DOVATO®, DTG/RPV), dolutegravir/lamivudine/tenofovir disoproxil fumarate (ACRIPTEGA/TELADOMYL/TENDOLA, TLD), dolutegravir/rilpivirine (JULUCA™, DTG/RPV), emtricitabine/tenofovir alafenamide (DESCOVY®, DVY), efavirenz (SUSTIVA®, STOCRIN®, EFV), efavirenz/emtricitabine/tenofovir disoproxil (ATRIPLA® ATR), efavirenz/lamivudine/tenofovir disoproxil fumarate (SYMFI™/SYMFI LO™, EFV/3TC/TDF), elvitegravir (VITEKTA®, EVG), elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (GENVOYA®, GEN), elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (STRIBILD®, STB), emtricitabine (EMTRIVA®, FTC), enfuvirtide (FUZEON®, T-20), entecavir (BARACLUDE®, ETV), etravirine (INTELENCE®, ETR), fosamprenavir calcium (LEXIVA®, FOS), fostemsavir (RUKOBIA, FTR), indinavir (CRIXIVAN®, IDV), lamivudine (EPIVIR®, 3TC), lamivudine/raltegravir (DUTREBIS™, DUT), lamivudine/tenofovir disoproxil fumarate (CIMDUO™, 3TC/TDF), lamivudine/zidovudine (COMBIVIR®, CBV), lenacapavir (SUNLENCA, LEN) lopinavir/ritonavir (KALETRA®, ALUVIA®, LPV/r), maraviroc (SELZENTRY®, CELSENTRI®, MVC), nelfinavir (VIRACEPT®, NFV), nevirapine (VIRAMUNE®, VIRAMUNE® XR™, NVP), raltegravir (ISENTRESS®, RAL), rilpivirine (EDURANT®, REKAMBYS®, CABENUVA®, RPV), rilpivirine/emtricitabine/tenofovir alafenamide (ODEFSEY®,ODE), rilpivirine/emtricitabine/tenofovir disoproxil (COMPLERA®, CPA; EVIPLERA®, EPA), ritonavir (NORVIR®, RTV), saquinavir (FORTOVASE®, SQV-SGC), saquinavir mesylate (INVIRASE®, SQV-HGC), stavudine (ZERIT®, d4T), telbivudine (SEBIVO®, TYZEKA®, LdT), tenofovir alafenamide (VEMLIDY®, TAF), tenofovir disoproxil fumarate (VIREAD®, TDF), tenofovir disoproxil fumarate/emtricitabine (TRUVADA®, TVD), tipranavir (APTIVUS®, TPV), zalcitabine (HIVID®, ddC), and zidovudine (RETROVIR®, ZDV).

ELIGIBILITY:
Eligibility Ages Eligible for Study: People of childbearing potential

Inclusion Criteria:

* Country of origin of report
* Documentation that the registry drug was taken during pregnancy
* Sufficient information to determine if the pregnancy is being prospectively or retrospectively registered
* Date the pregnancy was registered
* Source of report (patient or health care provider)
* Whether the pregnancy outcome is already known or delivery is still pending
* Timing of the prenatal exposure to the registry medication (no broader than which trimester)
* Sufficient patient identifier relevant to reporter to allow for follow-up
* Was patient involved in a study at the time of prenatal exposure
* Full reporter contact information (name, address, etc.)

Exclusion Criteria:

• People who were not exposed to registry medications during pregnancy

Ages: 12 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant people exposed to antiviral medications during pregnancy.
Sampling Method: Probability Sample
Enrollment: 24258 (Estimated)
Dates: Start 1989-01; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D Albano, PhD, MPH, Principal Investigator — Syneos Health
Locations (1):
- Registry Coordinating Center, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Vannappagari V, Albano JD, Koram N, Tilson H, Scheuerle AE, Napier MD. Prenatal exposure to zidovudine and risk for ventricular septal defects and congenital heart defects: data from the Antiretroviral Pregnancy Registry. Eur J Obstet Gynecol Reprod Biol. 2016 Feb;197:6-10. doi: 10.1016/j.ejogrb.2015.11.015. Epub 2015 Nov 24. PMID 26687320
- [Derived] Vannappagari V, Koram N, Albano J, Tilson H, Gee C. Association between in utero zidovudine exposure and nondefect adverse birth outcomes: analysis of prospectively collected data from the Antiretroviral Pregnancy Registry. BJOG. 2016 May;123(6):910-6. doi: 10.1111/1471-0528.13542. Epub 2015 Aug 12. PMID 26269220
- See also: Download: data forms to register patients, Semi-Annual Interim Report, product package inserts, organizational links, guidelines, bibliography — http://apregistry.com